CLINICAL TRIAL: NCT05107531
Title: Investigation of Gait, Foot Pressure Distribution and Balance in Parkinson's Patients With Motor Freezing
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Suleyman Korkusuz, Principal Investigator, Hacettepe University
Other Study IDs: GO21/777
Record Dates: First submitted 2021-10-18; First posted 2021-11-04 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Postural Balance; Parkinson's Disease; Gait Analysis; Kinematic Analysis; Motor Freezing; Spatio-Temporal Analysis; Foot Pressure Distribution
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Parkinson's Patients with Motor Freezing: Individuals with Parkinson's Disease with motor freezing were included in this group.
- Parkinson's Patients Without Motor Freeze: Individuals with Parkinson's Disease without motor freeze were included in this group.
- Healthy Controls: Healthy individuals who did not have any neurological problems that would affect gait were included.

SUMMARY:
Parkinson's disease is characterized by cardinal motor signs such as bradykinesia, tremor, rigidity and postural instability. In addition to these findings, motor freezing, gait disorders, posture disorders, decreased arm swings and loss of axial rotation are also seen. About 80% of the causes of falls in Parkinson's patients are due to postural instability and motor freezing, and patients' quality of life is significantly affected. In addition, gait disorders are common in advanced stages of Parkinson's Disease. Gait disorders decrease the quality of life by increasing the risk of falls, fractures and mortality. Therefore, the aim of this study is to observe the change in gait, foot pressure distribution and balance parameters of Parkinson's patients with and without motor deceleration compared to each other and healthy controls and to determine the relationship between these parameters.

DETAILED DESCRIPTION:
Parkinson's disease is characterized by basic motor symptoms such as bradykinesia, tremor, rigidity and postural instability. In addition to these findings, motor freezing, gait disorders, posture disorders, decreased arm swings and loss of axial rotation are also seen. Restrictions in balance, mobility and activities of daily living due to motor disorders seen in Parkinson's Disease and related disability, addiction and decrease in quality of life occur. Approximately 80% of the causes of falls in Parkinson's patients are due to postural instability and motor freezing, and the quality of life of patients is significantly affected. Also, gait disturbances are common in advanced stages of Parkinson's Disease. Gait disorders reduce the quality of life by increasing the risk of falls, fractures and death. Therefore, the aim of this study is to observe the changes in the gait, foot pressure distribution and balance parameters of Parkinson's patients with and without motor retardation compared to each other and to healthy controls, and to determine the relationship between these parameters.

This research is planned as two sub-work packages. Foot pressure distribution analysis and gait evaluation will be performed in the first sub-work package, and balance evaluation will be performed in the second sub-work package.

From the results of this research, 2 separate articles will be written that evaluate the balance and foot pressure distribution analysis and gait separately.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with idiopathic Parkinson's disease
* Healthy individuals who do not have musculoskeletal disease or any neurological disease that may affect assessments
* Being between 50-80 years old
* Volunteer to participate in the study
* Grade 2-3 on the Modified Hoehn-Yahr Scale
* To have a score above 24 in the Standardized Mini Mental Test

Exclusion Criteria:

* Having an additional neurological or psychiatric disease other than Parkinson's disease
* Uncontrollable dyskinesia or motor fluctuations
* Presence of postural hypotension, vision problems (not compensated by the correct lens) or vestibular disorders that may affect balance
* Presence of cardiopulmonary diseases that may affect gait
* Presence of orthopedic problems (such as fractures, osteoporosis, osteomyelitis) and inflammatory arthritis that may cause limitation of movement and affect gait and assessment

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parkinson's patients and healthy individuals who applied to Hacettepe University Neurology Clinic as voluntary participants will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-02-05 (Actual); Study Completion 2022-02-05 (Actual)

PRIMARY OUTCOMES:
E-LINK FP3 Force Plate | Baseline
  The system allows an accurate and objective assessment of the patient's ability to maintain postural stability on a static surface by measuring the symmetrical weight distribution in both the anterior-posterior and left-right axes. While the patient is standing on the force platform, a timed balance test is performed by the researcher to determine which direction the patient's balance has shifted.
KoreBalance Balance Evaluation System | Baseline
  KoreBalance is a balance assessment and training system designed with the latest technology. There is a variable air pressure pouch system and tilt sensor under the platform to monitor movements 360° horizontally and 20° vertically. There are dynamic and static balance tests in the device.
Functional Reach Test | Baseline
  The functional reach test is a dynamic test used to evaluate postural control. Participants are asked to reach forward through the ankle joint without moving their hips. Values less than 25.4 cm indicate an increased risk of falling.
Time Up and Go Test | Baseline
  The patient is asked to get up from the chair he is sitting in, walk three meters, turn around and sit again. At this time, the time is recorded. 10 seconds or less; It indicates that the patient walks independently, the risk of falling is low, and if it is longer than 30 seconds, it indicates the need for help from time to time and a high risk of falling.
Computerized Gait Assessment System (Zebris Rehawalk) | Baseline
  In addition to the spatiotemporal characteristics of gait such as gait speed, stride length, double stride length, stride width, cadence, stance and swing phase outputs, the pressure distribution measurement platform integrated into the system allows the measurement of dynamic foot pressure distribution. In addition, kinematic analysis of the gait can be made with the support of the camera in the system.

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale | Baseline
  It is used to evaluate the symptoms of the disease and the complications that develop due to treatment. In this scale, which consists of 4 parts, the scoring of each item is between 0-4 points. The increase in the total score reflects the increase in the severity of the symptoms.
Freezing of Gait Questionnaire | Baseline
  The scale is a scale that evaluates motor freezing in Parkinson's patients. It is questioned whether freezing occurs during activities such as walking and turning on the 6-item scale developed. In addition, in the presence of freezing, the severity, frequency and duration of freezing are recorded.

OTHER OUTCOMES:
Standardized Mini Mental Test | Baseline
  There are 19 items in this test, which consists of 5 main parts: orientation, recording memory, attention and calculation, recall and language. The total score of the test is evaluated out of 30 and 24 points are accepted as the threshold value for the diagnosis of mild dementia.
Modified Hoehn & Yahr Scale | Baseline
  It is the most frequently used scale to classify the progression stages of Parkinson's Disease. It is widely used for reasons such as being quite simple and being able to determine the motor and functional group of the patients. It performs the staging on the basis of the unilateral or bilateral status of the disease, and the effect on balance and gait. Progression in stages is associated with worsening motor and reduced quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Kadriye Armutlu, Prof. Dr., Study Chair — Hacettepe University; Süleyman Korkusuz, MSc, Principal Investigator — Hacettepe University; Emine Nur Demircan, MSc, Study Chair — Hacettepe University; Ayşenur Özcan, MSc, Study Chair — Hacettepe University; Büşra Seçkinoğulları, MSc, Study Chair — Hacettepe University; Gül Yalçın Çakmaklı, Assoc. Prof., Study Chair — Hacettepe University; Bülent Elibol, Prof. Dr., Study Chair — Hacettepe University; Ferdi Yavuz, Assoc. Prof., Study Chair
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schlenstedt C, Muthuraman M, Witt K, Weisser B, Fasano A, Deuschl G. Postural control and freezing of gait in Parkinson's disease. Parkinsonism Relat Disord. 2016 Mar;24:107-12. doi: 10.1016/j.parkreldis.2015.12.011. Epub 2015 Dec 18. PMID 26762797
- [Background] Mezzarobba S, Grassi M, Valentini R, Bernardis P. Postural control deficit during sit-to-walk in patients with Parkinson's disease and freezing of gait. Gait Posture. 2018 Mar;61:325-330. doi: 10.1016/j.gaitpost.2018.01.032. Epub 2018 Feb 2. PMID 29413805
- [Background] Bekkers EMJ, Dijkstra BW, Heremans E, Verschueren SMP, Bloem BR, Nieuwboer A. Balancing between the two: Are freezing of gait and postural instability in Parkinson's disease connected? Neurosci Biobehav Rev. 2018 Nov;94:113-125. doi: 10.1016/j.neubiorev.2018.08.008. Epub 2018 Aug 17. PMID 30125601
- [Background] Shah J, Pillai L, Williams DK, Doerhoff SM, Larson-Prior L, Garcia-Rill E, Virmani T. Increased foot strike variability in Parkinson's disease patients with freezing of gait. Parkinsonism Relat Disord. 2018 Aug;53:58-63. doi: 10.1016/j.parkreldis.2018.04.032. Epub 2018 May 1. PMID 29773512
- [Background] Chee R, Murphy A, Danoudis M, Georgiou-Karistianis N, Iansek R. Gait freezing in Parkinson's disease and the stride length sequence effect interaction. Brain. 2009 Aug;132(Pt 8):2151-60. doi: 10.1093/brain/awp053. Epub 2009 May 11. PMID 19433440
- [Background] Yang YR, Lee YY, Cheng SJ, Lin PY, Wang RY. Relationships between gait and dynamic balance in early Parkinson's disease. Gait Posture. 2008 May;27(4):611-5. doi: 10.1016/j.gaitpost.2007.08.003. Epub 2007 Sep 24. PMID 17890091